CLINICAL TRIAL: NCT03283462
Title: A Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Impact of a Daily Dose of AMAZ-02, a Food Derived Ingredient, for 4 Months on Skeletal Muscle Energetics and Function in Healthy Elderly
Brief Title: Bioenergetics and Muscle Function Improvement With AMAZ-02 in Elderly Skeletal Muscle (ENERGIZE Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: University of Washington (Other); Synteract, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 17.01.AMZ; 1178231 (Other: WIRB)
Record Dates: First submitted 2017-09-13; First posted 2017-09-14 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2020-10

CONDITIONS: Mitochondrial Function, Bioenergetics; Muscle Function; Aging

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mitopure (Active Comparator)
  Interventions: Dietary Supplement: Mitopure
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mitopure — Mitopure (Urolithin A) containing softgels
  Arms: Mitopure
Dietary Supplement: Placebo — Placebo containing softgels
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, single-center, placebo-controlled Phase 2 trial enrolling 66 healthy elderly subjects (33 placebo and 33 AMAZ-02 administration) who are ≥65 and ≤ 90 years of age with evidence of low mitochondrial function. AMAZ-02 or placebo will be orally administered for 4 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥65 and ≤90 years of age
2. Able to travel to and from the University of Washington and Fred Hutch Cancer Research Center (FHCRC)
3. Informed consent obtained
4. 6 minute walk distance of <550 meters
5. ATP max < 1mM /sec (in the hand FDI muscle)

Exclusion Criteria:

1. Subjects who have significant disease(s) or condition(s) which, in the opinion of the investigator, may put the subject at risk because of their participation in the trial or may influence either the results of the trial or the subject's ability to participate in the trial
2. Hospitalization within 3 months for major atherosclerotic events (defined as combined incidence of myocardial infarction, urgent target-vessel revascularization, coronary bypass surgery and stroke) and for any hospitalization within 2 months.
3. Have any metal implants in the right limbs, including non-MRI compatible metal stents, titanium pins/markers, etc.
4. Have an implanted cardiac pacemaker or other implanted non-MRI compatible cardiac device
5. Chronic, uncontrolled hypertension as judged by the Investigator (i.e., Baseline SBP >150 mm Hg, DBP >90 mm Hg) or a SBP > 150 mm Hg or DBP > 95 mm Hg at the time of screening or baseline. If the initial BP reading is above these values, the reading may be repeated one time within 20 minutes of the initial reading.
6. Body mass index <18 or >32 kg/m2
7. Severe chronic kidney disease requiring treatment with hemodialysis or peritoneal dialysis.
8. Additional laboratory abnormalities determined as clinically significant by the Investigator.
9. Clinically significant abnormalities on physical examination (as judged by the Investigator)
10. Clinically significant and chronic uncontrolled renal, hepatic, pulmonary, endocrine, neurologic disorders, bone, or gastrointestinal system dysfunction
11. History of seizures or epilepsy
12. History of serious mental illness as judged by the Investigator
13. Oral temperature >37.5°C at the time of the physical
14. Suspicion, or recent history, of alcohol or substance abuse or tobacco use
15. Subjects who in the opinion of the Investigator have a clinically significant abnormal 12-lead ECG during the screening period. Presence of atrial fibrillation, varying degrees of AV block, existence of a left bundle branch block, or evidence of previous myocardial infarction.
16. Subjects who are either unwilling to agree to refrain from using or are found to be using supplementary antioxidant vitamins (e.g., Coenzyme Q10, resveratrol, L-carnitine) from 7 days prior to dosing and throughout the treatment period
17. Subjects who are either unwilling to agree to refrain from using or are found to be using the following dietary restrictions (pomegranate juice, walnuts, pecans, strawberry, raspberry blackberry) from 7 days prior to dosing and throughout the treatment period
18. Are currently enrolled in a clinical trial involving an investigational product or non-approved use of a drug or device or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
19. Have participated, within the last 30 days from a clinical trial involving an investigational product. If the previous investigational product has a long half life, 3 months or 5 half-lives (whichever is longer) should have passed

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Change in 6 minute walking distance (6MWD) at the end of study intervention compared to baseline | 4 months
Percent change from baseline in ATP max (maximal ATP synthesis rate) in hand skeletal muscle (via Magnetic Resonance Spectroscopy) | 2, 4 months

SECONDARY OUTCOMES:
Percent change from baseline in contraction number during a hand muscle fatigue test | 2, 4 months
Percent change from baseline in ATP max (maximum ATP synthesis rate) in leg skeletal muscle (via MRS) | 4 months
Percent change from baseline in contraction number during a leg muscle fatigue test | 4 months
Change in Short Physical Performance Battery (SPPB) scores at the end of study intervention compared to baseline | 4 months
Change in exercise tolerance compared to baseline (via cycle ergometry) | 4 months
Change in hand grip strength at the end of study intervention compared to baseline | 4 months
Change in leg muscle strength (1-RM and 10-RM) at the end of study intervention compared to baseline | 4 months
Change in muscle size (cross-sectional area of the muscles) at the end of study intervention compared to baseline | 4 months
Change in mitochondrial function on muscle biopsy samples at the end of study intervention compared to baseline (via respirometry) | 4 months
Effect of AMAZ-02 on mitochondrial gene and protein expression in muscle tissue | 4 months
Effect of AMAZ-02 on plasma acylcarnitines | 4 months
Effect of AMAZ-02 on quality of life questionnaire (SF36) | 4 months
Change from baseline in plasma lipid profile | 4 months
Change from baseline in plasma for circulating biomarkers (myostatin, follistatin) | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: David Marcinek, PhD, Principal Investigator — University of Washington; Jose Garcia, MD, Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liu S, D'Amico D, Shankland E, Bhayana S, Garcia JM, Aebischer P, Rinsch C, Singh A, Marcinek DJ. Effect of Urolithin A Supplementation on Muscle Endurance and Mitochondrial Health in Older Adults: A Randomized Clinical Trial. JAMA Netw Open. 2022 Jan 4;5(1):e2144279. doi: 10.1001/jamanetworkopen.2021.44279. PMID 35050355